CLINICAL TRIAL: NCT00105378
Title: Effectiveness of EASYcare-based Geriatric Intermediate Care
Brief Title: Dutch EASYcare Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GEREASYEFF014-91-055; 014-91-055
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2007-08

CONDITIONS: Cognition Disorders; Mood Disorder; Gait Disorder, Neurologic; Malnutrition
Keywords: health care services research; frail elderly; intermediate care; patient centered care; comprehensive health care; geriatric nursing; Behavioral symptoms
MeSH Terms: conditions — Cognition Disorders; Mood Disorders; Gait Disorders, Neurologic; Malnutrition; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: Dutch EASYcare Study Geriatric Intermediate Care Programme

SUMMARY:
The purpose of this study is to study the effects of nursing home visits in independently living elderly people on their functional performance and health-related quality of life. The general practitioner (GP) can refer elderly people to this intervention model after identification of a problem in cognition, mood, behavior, mobility, or nutrition. A specialist geriatric nurse visits the patients at home up to six times and coaches the patient in cooperation with the GP and geriatrician.

DETAILED DESCRIPTION:
General practitioners (GPs) in the Western world have to anticipate the increasing age and health care demands of their patients. A considerable proportion of those older patients have reduced functional status and quality of life, which may affect their feelings of autonomy and ability to live independently. Even with considerable disability, most patients prefer to stay at home. Because of their complex clinical presentations and needs, these patients require a special approach to their evaluation and care.

Intermediate care is a possible answer to these changing demands, although the efficacy of these programs is a subject of vivid debate.

With the Dutch Geriatric Intermediate Care Programme (DGIP) we developed an Intermediate Care model to study efficacy aspects of problem based intermediate care. DGIP is an intermediate care program in which the GP refers elderly patients with a problem in cognition, mood, behavior, mobility, and nutrition. A geriatric specialist nurse applies a guideline based intervention in a maximum of six visits during a maximum of three months. The nurse starts the intervention with the application of the EASYcare instrument for geriatric screening. The EASYcare instrument assesses (instrumental) activities of daily life, cognition, mood, and includes a goal setting item. During the intervention the nurse regularly consults the referring GP and a geriatrician.

Objectives

* To determine the effects of the Dutch EASYcare Study Geriatric Intermediate care Programme compared to regular medical care in improving health related quality of life in independently living elderly persons and their informal caregivers who contact the GP with one of a variety of geriatric problems.
* To determine the costs of the Dutch EASYcare Study Geriatric Intermediate care Programme.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age and over
* The patient lives independently or in a home for the aged
* The patient has a health problem that was recently presented to the GP by the patient or informal caregiver
* The request for help is related to the following problem fields: cognitive disorders, behavioral and psychological symptoms of dementia, mood disorders, mobility disorders and falling, or malnutrition
* The patient/informal caregiver and GP have determined a goal they want to achieve
* Fulfill one or more of these criteria: MMSE (Mini Mental State Examination) equal to or less than 26, GARS (Groningen Activity Restriction Scale) equal to or greater than 25 or MOS-20/subscale mental health equal to or less than 75

Exclusion Criteria:

* The problem or request for help has an acute nature, urging for action (medical or otherwise) within less than one week
* The problem or request for help is merely a medical diagnostic issue, urging for action only physicians (GP or specialist) can offer
* MMSE < 20 or proved moderate to severe dementia (Clinical Dementia Rating scale [CDR] > 1, 0) and no informal caregiver (no informal caregiver is defined as: no informal caregiver who meets the patient for at least once a week on average)
* The patient receives other forms of intermediate care or health care from a social worker or community-based geriatrician
* The patient is already on the waiting list for a nursing home because of the problem the patient is presented with in our study
* Predicted prognosis < 6 months because of terminal illness

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 155 (Actual)
Dates: Start 2003-04; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Functional performance (independent) activities of daily living measured using Groningen Activity Restriction Scale | 3 months
Mental health using subscale mental health MOS-20 | 3 months
Informal caregiver burden using Zarit Burden Interview | 3 months

SECONDARY OUTCOMES:
Type of residence (independent, home for the elderly, nursing home) | 3 months
Cost effectiveness | 6 months
Mobility using Timed Up and Go test | 3 months
Overall health related Quality of life using MOS-20 | 3 months
Well-being using Cantril Self-anchoring ladder and Dementia Quality of Life | 3 months
Cognition using Mini Mental State Examination | 6 months
Social functioning using Loneliness scale de Jong-Gierveld | 3 months
Subjective treatment effects using Patient Enablement Instrument | 3 months
Mortality | within a period of maximum two years
Time spent on care by informal caregiver | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcel G. Olde Rikkert, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Borm GF, Melis RJ, Teerenstra S, Peer PG. Pseudo cluster randomization: a treatment allocation method to minimize contamination and selection bias. Stat Med. 2005 Dec 15;24(23):3535-47. doi: 10.1002/sim.2200. PMID 16007575
- [Background] Richardson J. The Easy-Care assessment system and its appropriateness for older people. Nurs Older People. 2001 Oct;13(7):17-9. doi: 10.7748/nop.13.7.17.s15. No abstract available. PMID 12008559
- [Derived] Melis RJ, Adang E, Teerenstra S, van Eijken MI, Wimo A, van Achterberg T, van de Lisdonk EH, Rikkert MG. Cost-effectiveness of a multidisciplinary intervention model for community-dwelling frail older people. J Gerontol A Biol Sci Med Sci. 2008 Mar;63(3):275-82. doi: 10.1093/gerona/63.3.275. PMID 18375876